CLINICAL TRIAL: NCT04040296
Title: Personalized Recommendations for Acute Kidney Injury (AKI) Care Using a Kidney Action Team: A Randomized Trial
Brief Title: Personalized Recommendations for Acute Kidney Injury (AKI) Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2000026203
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Results first posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Kidney Action Team Recommendations will not be delivered to the primary care teams of randomized patients.
- Kidney Action Team Recommendations (Experimental): Recommendations made by the Kidney Action Team will be delivered to the patient's primary care team within 2 hours of AKI detection.
  Interventions: Other: Kidney Action Team Recommendations

INTERVENTIONS:
Other: Kidney Action Team Recommendations — Upon review of the patient's medical information, the Kidney Action Team will create personalized recommendations that will be delivered to the patient's primary care team via a specialized note in the electronic medical record system within 2 hours of AKI detection. The attending of record will be identified as a cosigner to ensure that a member of the care team is made aware of the note's presence.
  Arms: Kidney Action Team Recommendations

SUMMARY:
This is a randomized clinical trial of a "Kidney Action Team", which will provide timely, personalized recommendations for the diagnosis and initial treatment of hospitalized patients with Acute Kidney Injury (AKI).

DETAILED DESCRIPTION:
Acute Kidney Injury (AKI), defined as an abrupt loss in kidney function, is common, occurring in 5-20% of hospitalized patients, and carries a significant and independent risk of inpatient mortality. International guidelines for the treatment of AKI focus on "best practices" that include appropriate management of drug dosing, the avoidance of kidney-toxic exposures, and careful assessment of fluid and electrolyte balance. Early nephrologist involvement may also improve outcomes in AKI. However, AKI, which is often asymptomatic, is frequently overlooked in a variety of hospital settings and many "best practices" occur infrequently and inconsistently.

The investigators previously conducted a randomized clinical trial testing the efficacy of electronic alerts for AKI, randomizing patients with AKI to usual care, or to an alert group in which a single alert was sent to the patient's primary provider. The study demonstrated clinical equipoise regarding the effectiveness of such alerting, as there was no improvement in the rates of AKI progression, dialysis or mortality among those in the alert group.

Rather than simply making providers aware of AKI, it may be beneficial to provide them with actionable items to increase recognition and rate of best practices. Further, because of the heterogeneous nature of AKI, personalized recommendations tailored to individual patients that are delivered directly to the patient care team may improve AKI outcomes. The aim of this study is to determine, through a single-blind, parallel group, randomized controlled multicenter clinical trial, if personalized recommendations, as delivered by a Kidney Action Team, for the work-up and treatment of AKI will improve patient outcomes. The Kidney Action team will serve as a centralized, remote monitoring service and will consist of a group of highly trained individuals, including an advanced practitioner, a pharmacist and a board-certified nephrologist, dedicated to reviewing enrolled patient's charts and providing recommendations for patient diagnosis and initial work up and care within 60 minutes of AKI onset. Recommendations will span five domains of care, including diagnostic workup, acid/base management, electrolyte management, hemodynamic management, and medication management.

Using the Kidney Disease: Improve Global Outcomes creatinine criteria, inpatients in sites of the Yale New Haven Health System and of the John Hopkins University Health System who develop AKI during the course of their hospitalization will be randomized to either receive usual care, or to an active intervention group in which the recommendations of the Kidney Action Team are delivered to the patient's primary care team in the form of a structured note in the electronic health record to be cosigned by the attending of record. The primary clinical outcome will be a composite of AKI progression, dialysis and death at 14 days post-randomization. The primary process outcome will be the percent of recommendations made that are enacted within 24 hours after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years admitted to a participating hospital (six hospitals in the Yale New Haven Health system and two hospitals of the John Hopkins University Health system)
2. Stage 1 Acute Kidney Injury as defined by KDIGO creatinine criteria:

   * 0.3 mg/dl increase in inpatient serum creatine over 48 hours OR
   * 50% relative increase in inpatient serum creatinine over 168 hours

Exclusion Criteria:

1. Admission to hospice service or comfort measures only order
2. Recipient of a solid organ transplant
3. Immediate dialytic indication determined by the following:

   * serum K >/= 7
   * arterial pH < 7.15
   * BUN > 150 mg/dL
   * acute ingestion of dialyzable toxins
   * refractory volume overload

   Patients who meet any of these critical values will not be enrolled in the trial and the Kidney Action Team will directly notify the treating team.
4. Pre-existing CKD stage V or End Stage Kidney Disease
5. Initial hospital creatinine > 4.0 mg/dl
6. Patients who have been seen by nephrology or already have a nephrology consult
7. Status post-nephrectomy (partial or radical) during index admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4003 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis P Wilson, Principal Investigator — Yale Univerisity
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified aggregate data for the primary and secondary outcomes will be made available.
Supporting Information: Study Protocol
Time Frame: Data will be made available within one year of completion.

REFERENCES:
- [Background] Wilson FP, Shashaty M, Testani J, Aqeel I, Borovskiy Y, Ellenberg SS, Feldman HI, Fernandez H, Gitelman Y, Lin J, Negoianu D, Parikh CR, Reese PP, Urbani R, Fuchs B. Automated, electronic alerts for acute kidney injury: a single-blind, parallel-group, randomised controlled trial. Lancet. 2015 May 16;385(9981):1966-74. doi: 10.1016/S0140-6736(15)60266-5. Epub 2015 Feb 26. PMID 25726515
- [Derived] Aklilu AM, Menez S, Baker ML, Brown D, Dircksen KK, Dunkley KA, Gaviria SC, Farrokh S, Faulkner SC, Jones C, Kadhim BA, Le D, Li F, Makhijani A, Martin M, Moledina DG, Coronel-Moreno C, O'Connor KD, Shelton K, Shvets K, Srialluri N, Tan JW, Testani JM, Corona-Villalobos CP, Yamamoto Y, Parikh CR, Wilson FP; KAT-AKI Team. Early, Individualized Recommendations for Hospitalized Patients With Acute Kidney Injury: A Randomized Clinical Trial. JAMA. 2024 Dec 24;332(24):2081-2090. doi: 10.1001/jama.2024.22718. PMID 39454050
- [Derived] Aklilu AM, O'Connor KD, Martin M, Yamamoto Y, Coronel-Moreno C, Shvets K, Jones C, Kadhim B, Corona-Villalobos CP, Baker ML, Tan J, Freeman N, Groener M, Menez S, Brown D, Culli SE, Lindsley J, Orias M, Parikh C, Smith A, Sundararajan A, Wilson FP. Personalised recommendations for hospitalised patients with Acute Kidney Injury using a Kidney Action Team (KAT-AKI): protocol and early data of a randomised controlled trial. BMJ Open. 2023 Apr 17;13(4):e071968. doi: 10.1136/bmjopen-2023-071968. PMID 37068906

RESULTS

PARTICIPANT FLOW:
Groups:
- Kidney Action Team Recommendations: Recommendations made by the Kidney Action Team will be delivered to the patient's primary care team within 2 hours of AKI development.
  Kidney Action Team Recommendations: Upon review of the patient's medical information, the Kidney Action Team will create personalized recommendations that will be delivered to the patient's primary care team via a specialized note in the electronic medical record system within 2 hours of AKI development. The attending of record will be identified as a cosigner to ensure that a member of the care team is made aware of the note's presence.
Period: Overall Study
Arm/Group | Usual Care | Kidney Action Team Recommendations
Started | 2004 | 1999
Completed | 2004 | 1999
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Kidney Action Team Recommendations | Total
Number analyzed (Participants) | 2004 | 1999 | 4003
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 71.8 [60.6 to 81.3] | 71.9 [60.3 to 81.3] | 71.9 [60.5 to 81.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 964 | 910 | 1874
  Male | 1040 | 1089 | 2129
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 467 | 464 | 931
  White | 1336 | 1325 | 2661
  Other | 201 | 210 | 411
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic ethnicity, n (%) | 170 | 171 | 341
Hypertension, n (%) [Count of Participants; unit: Participants] | 1645 | 1602 | 3247
Diabetes mellitus, n (%) [Count of Participants; unit: Participants] | 957 | 927 | 1884
Congestive Heart Failure, n (%) [Count of Participants; unit: Participants] | 913 | 872 | 1785
Chronic Kidney Disease, n (%) [Count of Participants; unit: Participants] | 825 | 840 | 1665
Atrial fibrillation, n (%) [Count of Participants; unit: Participants] | 666 | 601 | 1267
Chronic obstructive pulmonary disease, n (%) [Count of Participants; unit: Participants] | 630 | 577 | 1207
Cirrhosis, n (%) [Count of Participants; unit: Participants] | 135 | 135 | 270
Malignancy, n (%) [Count of Participants; unit: Participants] | 110 | 120 | 230
Elixhauser comorbidity score [Median (Inter-Quartile Range); unit: units on a scale] — A comorbidity index score used to quantify comorbid conditions based on the presence of 31 pre-existing conditions (using ICD diagnosis codes) scored as present or not. Single scores range 0 from to 31, with higher scores predicting higher in-hospital mortality rates.
  units on a scale | 8 [4 to 12] | 7 [4 to 12] | 8 [4 to 12]
Serum creatinine, median (IQR), mg.dL [Median (Inter-Quartile Range); unit: mg/dL] | 1.17 [.9 to 1.59] | 1.19 [.9 to 1.55] | 1.18 [.9 to 1.57]
Estimated glomerular filtration rate, median (IQR), mL/min [Median (Inter-Quartile Range); unit: mL/min] | 57.7 [40.3 to 84.7] | 58.2 [40.3 to 82.6] | 57.9 [40.3 to 83.8]
Hospital site, n (%) [Count of Participants; unit: Participants]
  Yale | 1602 | 1598 | 3200
  John Hopkins | 402 | 401 | 803
Hospital service [Count of Participants; unit: Participants]
  General medical floor | 1014 | 983 | 1997
  ICU/SDU units | 404 | 382 | 786
  Surgical floor | 327 | 340 | 667
  Specialist medical floor | 259 | 294 | 553
Hospital service- General medical floor under hospitalist care, n (%) [Count of Participants; unit: Participants] | 716 | 713 | 1429
Hospital service- General medical floor under teaching medical team, n (%) [Count of Participants; unit: Participants] | 298 | 270 | 568
mSOFA, median (IQR) [Median (Inter-Quartile Range); unit: units on a scale] — The Modified Sequential Organ Failure Assessment score, used to predict mortality in critically ill patients. Each of five organ systems is scored on a scale from 0-4, with 4 indicating the highest dysfunction. The scores are summed to total 0 to 20, with a mSOFA score of 20 indicating highest dysfunction.
  units on a scale | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]
AKI stage at diagnosis [Count of Participants; unit: Participants] — AKI staged using Kidney Outcomes Improving Global Outcomes (KDIGO) criteria, whereby stage 1 is defined as an increase in serum creatinine of 0.3mg/dL over 48 hours or a relative increase of 50% from baseline over 7 days, stage 2 is defined by an increase by 2 to < 3 times from the lowest creatinine within the prior 7 days., and stage 3 is defined by an increase of > 3 times from the lowest within the prior 7 days or requirement of dialysis. A higher stage indicates worsening disease state and worse outcomes.
  Participants
    0 | 20 | 19 | 39
    1 | 1823 | 1825 | 3648
    2 | 139 | 132 | 271
    3 | 22 | 23 | 45
sCR, mg/dL [Median (Inter-Quartile Range); unit: mg/dL] | 1.5 [1.21 to 1.95] | 1.52 [1.26 to 1.97] | 1.5 [1.23 to 1.96]
BUN, md/dL [Median (Inter-Quartile Range); unit: mg/dL] | 28.5 [20 to 40] | 29 [20 to 40] | 29 [20 to 40]
Potassium, mEq/L [Median (Inter-Quartile Range); unit: mEq/L] | 4.2 [3.8 to 4.6] | 4.2 [3.8 to 4.6] | 4.2 [3.8 to 4.6]
Bicarbonate, mEq/L [Median (Inter-Quartile Range); unit: mEq/L] | 24 [21 to 27] | 24 [21 to 27] | 24 [21 to 27]
White blood cell count [Median (Inter-Quartile Range); unit: x10^3 cells/uL] | 9.1 [6.8 to 13] | 9.4 [6.7 to 13.1] | 9.2 [6.8 to 13.1]
Hemoglobin, g/dL [Median (Inter-Quartile Range); unit: g/dL] | 10.6 [8.9 to 12.4] | 10.5 [8.9 to 12.4] | 10.6 [8.9 to 12.4]
Platelet count [Median (Inter-Quartile Range); unit: x10^3 cells/uL] | 212 [155 to 281] | 211 [153 to 282] | 212 [153 to 281]
Exposures [Count of Participants; unit: Participants]
  Antibiotics | 533 | 554 | 1087
  Contrast | 407 | 440 | 847
  NSAIDs | 176 | 195 | 371
  Sustained hypotension | 187 | 186 | 373
  Vasopressor | 11 | 17 | 28
Recommendations category [Count of Participants; unit: Participants] — Recommendations were made upon enrollment within 1-2 hours of AKI detection and prior to randomization and are as such considered part of the exposure, rather than an outcome.
  Participants
    General | 1931 | 1920 | 3851
    Volume | 1589 | 1606 | 3195
    Potassium | 315 | 307 | 622
    Acid-base | 208 | 200 | 408
    Renal consult | 34 | 36 | 70
    Medication | 1114 | 1069 | 2183
Recommendation count, median (IQR) [Median (Inter-Quartile Range); unit: number of recommendations] — Recommendations were made upon enrollment within 1-2 hours of AKI detection and prior to randomization and are as such considered part of the exposure, rather than an outcome.
  number of recommendations | 3 [2 to 5] | 3 [2 to 5] | 3 [2 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Composite Outcome Showing the Percentage of Participants With Any One of the Following: Progression of AKI, Inpatient Dialysis, or Inpatient Death
Description: Progression of AKI is defined by an increase in KDIGO creatinine stage from that present at the time of randomization.
  Dialysis is defined by the receipt of hemodialysis, continuous renal replacement therapy or peritoneal dialysis. Isolated ultrafiltration treatments (for the purpose of volume removal) will not be included.
  Mortality will be determined from hospital administrative records.
  The rates of the primary outcome will be compared between the study arms using the Cochrane-Mantel-Haenszel chi-square test, accounting for stratification by hospital.
Time Frame: 14 days post randomization or at hospital discharge, whichever comes first
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Kidney Action Team Recommendations
Number analyzed (Participants) | 2004 | 1999
Participants | 369 | 395
Statistical Analysis 1: Comparison: Usual Care vs Kidney Action Team Recommendations; Test type: Superiority; p = 0.28, Cochran-Mantel-Haenszel; Difference in percentage = 1.4, 95% CI 2-sided [-1.1 to 3.8] — Difference between arms in the percentage of subjects with the primary outcome within 14 days of randomization

2. Secondary Outcome: Percentage of Recommendations Implemented by the Primary Care Team
Description: The AKI Response Team will make recommendations for all randomized patients in both the control group and the intervention group, however, recommendations will only be delivered to the primary care teams of patients in the intervention group. In this way, we can compare the percentage of recommendations that were followed by primary care teams across both groups. This outcome will be assessed by averaging the proportion of recommendations followed within 24 hours between the two study arms using the Van Elteren test to account for stratification by hospital.
Time Frame: 24 hours after randomization
Measure: Number; unit: Number of recommendations
Arm/Group | Usual Care | Kidney Action Team Recommendations
Number analyzed (Participants) | 2004 | 1999
Number of recommendations
  Recommendations completed | 1766 | 2459
  Recommendations made | 7269 | 7270
Statistical Analysis 1: Comparison: Usual Care vs Kidney Action Team Recommendations; Proportions were compared using Cochrane-Mantel Haenszel χ2 test, accounting for stratification by hospital site; Test type: Superiority; p < .001, Van Elteren test; Difference in percentage = 9.5, 95% CI 2-sided [8.1 to 11] — Difference between arms in the percentage of implemented recommendations with 24 hours of randomization

3. Secondary Outcome: Percentage of Patients With Progression of Acute Kidney Injury
Description: Percentage of patients who progressed from stage 1 to stage 2 or 3 or from stage 2 to stage 3 (based on changes in creatinine) within 14 days of randomization
Time Frame: Assessed from time of randomization to time of AKI progression (within 14 days post randomization)
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Kidney Action Team Recommendations
Number analyzed (Participants) | 2004 | 1999
Participants | 261 | 270
Statistical Analysis 1: Comparison: Usual Care vs Kidney Action Team Recommendations; Proportions were compared using Cochrane-Mantel Haenszel χ2 test, accounting for stratification by hospital site; Test type: Superiority; p = .65, Van Elteren test; Difference in percentage = .5, 95% CI 2-sided [-1.6 to 2.6] — Difference between arms in the percentage of subjects with AKI progression within 14 days of randomization

4. Secondary Outcome: Percentage of Patients Who Receive Inpatient Dialysis
Description: Percentage of patients who receive hemodialysis, continuous renal replacement, or peritoneal dialysis during index hospitalization within 14 days of randomization
Time Frame: Assessed from time of randomization to time of receipt of inpatient dialysis (within 14 days post randomization)
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Kidney Action Team Recommendations
Number analyzed (Participants) | 2004 | 1999
Participants | 30 | 31
Statistical Analysis 1: Comparison: Usual Care vs Kidney Action Team Recommendations; Proportions were compared using Cochrane-Mantel Haenszel χ2 test, accounting for stratification by hospital site; Test type: Superiority; p = .89, Van Elteren test; Difference in percentage = .1, 95% CI 2-sided [-.7 to .8] — Difference between arms in the percentage of subjects who received inpatient dialysis within 14 days of randomization

5. Secondary Outcome: Percentage of Inpatient Mortality
Description: Proportion of patients who expire within 14 days of randomization
Time Frame: Assessed from time of randomization to date of death from any cause, within 14 days of randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Kidney Action Team Recommendations
Number analyzed (Participants) | 2004 | 1999
Participants | 185 | 191
Statistical Analysis 1: Comparison: Usual Care vs Kidney Action Team Recommendations; Proportions were compared using Cochrane-Mantel Haenszel χ2 test, accounting for stratification by hospital site; Test type: Superiority; p = .72, Van Elteren test; Difference in percentage = .4, 95% CI 2-sided [-1.5 to 2.1] — Difference between arms in the percentage of subjects with inpatient mortality within 14 days of randomization

6. Secondary Outcome: Percent of Patients Who Receive a Kidney Consult Within 14 Days
Description: Percent of participants receiving a kidney consult within 14 days of randomization
Time Frame: Assessed from the time of randomization to time of first kidney consult (within 14 days post-randomization)
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Kidney Action Team Recommendations
Number analyzed (Participants) | 2004 | 1999
Participants | 284 | 321
Statistical Analysis 1: Comparison: Usual Care vs Kidney Action Team Recommendations; Proportions were compared using Cochrane-Mantel Haenszel χ2 test, accounting for stratification by hospital site; Test type: Superiority; p = .31, Van Elteren test; Difference in percentage = 1.9, 95% CI 2-sided [-.3 to 4.1] — Difference between arms in the percentage of subjects who received a kidney consult within 14 days of randomization

7. Secondary Outcome: Percent of Patients Who Are Discharged to Hospice Care 14 Days
Description: Percent of participants discharged to hospice within 14 days of randomization
Time Frame: Assessed from the time of randomization to time discharge to hospice (within 14 days post-randomization)
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Kidney Action Team Recommendations
Number analyzed (Participants) | 2004 | 1999
Participants | 106 | 87
Statistical Analysis 1: Comparison: Usual Care vs Kidney Action Team Recommendations; Proportions were compared using Cochrane-Mantel Haenszel χ2 test, accounting for stratification by hospital site; Test type: Superiority; p = .17, Van Elteren test; Difference in percentage = -.9, 95% CI 2-sided [-2.3 to .4] — Difference between arms in the percentage of subjects discharged to hospice care within 14 days of randomization

ADVERSE EVENTS:
Time Frame: Adverse events were assessed unsystematically by provider reporting throughout the trial and until study completion, to be reviewed by the internal team and external DSMB. The study lasted 2 years and 4 months, with each subject enrolled for 14 days in which adverse events could be reported.
Groups:
- Kidney Action Team Recommendations: Recommendations made by the Kidney Action Team will be delivered to the patient's primary care team within 60 minutes of AKI development.
  Kidney Action Team Recommendations: Upon review of the patient's medical information, the Kidney Action Team will create personalized recommendations that will be delivered to the patient's primary care team via a specialized note in the electronic medical record system within 60 minutes of AKI development. The attending of record will be identified as a cosigner to ensure that a member of the care team is made aware of the note's presence.
Arm/Group | Usual Care | Kidney Action Team Recommendations
All-Cause Mortality (participants affected / at risk) | 185/2004 | 191/1999
Serious Adverse Events (participants affected / at risk) | 0/2004 | 0/1999
Other Adverse Events (participants affected / at risk) | 0/2004 | 0/1999

LIMITATIONS AND CAVEATS:
Timely notice, adherence and implementation of recommendations by providers was not guaranteed. Limited windows of time for enrollment may have introduced bias that affected outcomes. Given the bundled nature of the recommendations, the unique effects of a given recommendation could not be determined. Finally, though the structured recommendation form was broad and included an option for free-text recommendations, it is possible that other recommendations may have led to different effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT04040296/Prot_SAP_000.pdf